CLINICAL TRIAL: NCT00178087
Title: Pathways Linking Late-Life Depression to MCI & Dementia
Brief Title: Determining Changes in Brain Structure Associated With Symptoms of Late-life Depression
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Meryl Butters, Associate Professor, University of Pittsburgh
Other Study IDs: R01MH072947 (NIH); R01MH072947 (NIH); 9512127; DATR A4-GPT
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Late-Life Depression
Keywords: late-life depression; mild cognitive impairment; dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will determine the changes in brain structure and function that are responsible for mood and cognition changes that are sometimes associated with late-life depression.

DETAILED DESCRIPTION:
The goal of this research study is to investigate the relationships among late-life depression (LLD), cognitive impairment and progressive neurodegeneration. The guiding hypothesis is that LLD patients have evolving cognitive impairments as a consequence of distinct underlying neuropathological changes, which frequently are expressed as Mild Cognitive Impairment (MCI). These neuropathological and cognitive changes are risk modifiers, lowering brain reserve capacity, and in turn, increasing risk of developing Alzheimer's Disease (AD). In order to pursue this goal we will enroll LLD, MCI, and normal control subjects to enrich our existing cohort to include a total of 150 elderly, non-demented, non-depressed subjects, 60 non-depressed MCI subjects and 270 LLD subjects. Using the joint infrastructure of the University of Pittsburgh's Advanced Center for Intervention and Services Research for Late-Life Mood Disorders and the Alzheimer's Disease Research Center, we will complete a detailed neurobehavioral evaluation, including clinical, neuropsychological, neuroimaging and biological markers, using these data to evaluate the factors associated with the development of MCI or dementia. Subjects will be studied annually for at least three years, allowing us to use longitudinal data to evaluate a series of linked hypotheses that postulate the pathways by which elderly, depressed patients develop cognitive impairment, and which may lead some to develop dementia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a mood disorder

Exclusion Criteria:

* Major acute medical illnesses or injuries known to have significant direct effects on cognitive functioning (e.g., metastatic cancer, multiple sclerosis, traumatic brain injury).
* Uncorrectable sensory handicap (e.g., blindness), because they are unable to complete the cognitive test battery.
* Exclusion criteria for MR scans include: cardiac pacemaker, aneurysm clip, cochlear implant, pregnancy, IUD, shrapnel, history of metal fragments in the eye, neurostimulators, weight of 250 lbs. or more, or claustrophobia.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 150 elderly, non-demented, non-depressed subjects, 60 non-depressed mild cognitive impairment subjects and 270 late-life depression subjects
Sampling Method: Non-Probability Sample
Enrollment: 331 (Actual)
Dates: Start 2005-08; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Changes in performance on a broad-based Neuropsychological Test Battery | 3 years
  Changes in z-scores of the language, visuospatial, attention, memory and executive cognitive domains

CONTACTS AND LOCATIONS:
Overall Officials: Meryl A. Butters, Ph.D., Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - UPMC Late-Life Evaluation and Treatment Center, Pittsburgh, Pennsylvania
  - UPMC Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Butters MA, Whyte EM, Nebes RD, Begley AE, Dew MA, Mulsant BH, Zmuda MD, Bhalla R, Meltzer CC, Pollock BG, Reynolds CF 3rd, Becker JT. The nature and determinants of neuropsychological functioning in late-life depression. Arch Gen Psychiatry. 2004 Jun;61(6):587-95. doi: 10.1001/archpsyc.61.6.587. PMID 15184238
- [Background] Butters MA, Sweet RA, Mulsant BH, Ilyas Kamboh M, Pollock BG, Begley AE, Reynolds CF 3rd, DeKosky ST. APOE is associated with age-of-onset, but not cognitive functioning, in late-life depression. Int J Geriatr Psychiatry. 2003 Dec;18(12):1075-81. doi: 10.1002/gps.1006. PMID 14677138
- [Background] Butters MA, Becker JT, Nebes RD, Zmuda MD, Mulsant BH, Pollock BG, Reynolds CF 3rd. Changes in cognitive functioning following treatment of late-life depression. Am J Psychiatry. 2000 Dec;157(12):1949-54. doi: 10.1176/appi.ajp.157.12.1949. PMID 11097959
- [Background] Bell-McGinty S, Butters MA, Meltzer CC, Greer PJ, Reynolds CF 3rd, Becker JT. Brain morphometric abnormalities in geriatric depression: long-term neurobiological effects of illness duration. Am J Psychiatry. 2002 Aug;159(8):1424-7. doi: 10.1176/appi.ajp.159.8.1424. PMID 12153839
- [Background] Nebes RD, Pollock BG, Houck PR, Butters MA, Mulsant BH, Zmuda MD, Reynolds CF 3rd. Persistence of cognitive impairment in geriatric patients following antidepressant treatment: a randomized, double-blind clinical trial with nortriptyline and paroxetine. J Psychiatr Res. 2003 Mar-Apr;37(2):99-108. doi: 10.1016/s0022-3956(02)00085-7. PMID 12842163
- [Background] Sweet RA, Hamilton RL, Butters MA, Mulsant BH, Pollock BG, Lewis DA, Lopez OL, DeKosky ST, Reynolds CF 3rd. Neuropathologic correlates of late-onset major depression. Neuropsychopharmacology. 2004 Dec;29(12):2242-50. doi: 10.1038/sj.npp.1300554. PMID 15354182
- [Background] Lopez OL, Jagust WJ, DeKosky ST, Becker JT, Fitzpatrick A, Dulberg C, Breitner J, Lyketsos C, Jones B, Kawas C, Carlson M, Kuller LH. Prevalence and classification of mild cognitive impairment in the Cardiovascular Health Study Cognition Study: part 1. Arch Neurol. 2003 Oct;60(10):1385-9. doi: 10.1001/archneur.60.10.1385. PMID 14568808
- [Background] Lopez OL, Jagust WJ, Dulberg C, Becker JT, DeKosky ST, Fitzpatrick A, Breitner J, Lyketsos C, Jones B, Kawas C, Carlson M, Kuller LH. Risk factors for mild cognitive impairment in the Cardiovascular Health Study Cognition Study: part 2. Arch Neurol. 2003 Oct;60(10):1394-9. doi: 10.1001/archneur.60.10.1394. PMID 14568809
- [Background] Thompson PM, Hayashi KM, de Zubicaray G, Janke AL, Rose SE, Semple J, Herman D, Hong MS, Dittmer SS, Doddrell DM, Toga AW. Dynamics of gray matter loss in Alzheimer's disease. J Neurosci. 2003 Feb 1;23(3):994-1005. doi: 10.1523/JNEUROSCI.23-03-00994.2003. PMID 12574429
- [Background] Ballmaier M, Toga AW, Blanton RE, Sowell ER, Lavretsky H, Peterson J, Pham D, Kumar A. Anterior cingulate, gyrus rectus, and orbitofrontal abnormalities in elderly depressed patients: an MRI-based parcellation of the prefrontal cortex. Am J Psychiatry. 2004 Jan;161(1):99-108. doi: 10.1176/appi.ajp.161.1.99. PMID 14702257
- See also: Related Info — http://www.wpic.pitt.edu/research/depr/